CLINICAL TRIAL: NCT00168246
Title: A Cross-Sectional Study of HIV-Related Neurological Disorders in Ten Countries of the Asia Pacific Region
Brief Title: Determining the Prevalence of HIV-Related Neurological Disorders in the Asia Pacific
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Collaborators: The Alfred (Other); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Other Study IDs: 77/05
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2007-02-27 (Estimated); Status verified 2007-02

CONDITIONS: HIV Infections; HIV Related Neurological Diseases
Keywords: HIV
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Natural History | Time Perspective: Other

SUMMARY:
This study will determine the prevalence of HIV-related neurological disorders in the countries of the Asia-Pacific Region.

DETAILED DESCRIPTION:
This a cross-sectional study to determine the prevalence of HIV-related Neurological Disorders in the countries of the Asia-Pacific Region. Researchers will visit each country site for a period of 2-3 weeks and work with local investigators. Outpatients will be evaluated once-only for the presence of HIV-related symptomatic peripheral neuropathy and HIV-related Neurocognitive Impairment. Inpatients at the sites will be evaluated once-only for the presence of HIV dementia, cerebral toxoplasmosis, cerebral tuberculosis, cryptococcal meningitis, lymphoma, PML and CMV encephalitis.

The Primary outcomes are:

1. To determine the prevalence of HIV-related neurocognitive impairment and ADC at the APNAC-10 sites
2. To determine the prevalence of symptomatic peripheral sensory neuropathy at the APNAC-10 sites
3. To determine the prevalence of central nervous system opportunistic infections and tumours at the APNAC-10 sites

The secondary outcomes are:

To determine the degree of cognitive impairment in patients presenting with HIV-related cognitive impairment at the APNAC-10 sites

* To determine the CD4 cell counts, HIV viral loads HIV viral loads and prior AIDS defining illnesses (ADIs) of patients presenting with HIV-related neurocognitive impairment and ADC at the APNAC-10 sites
* To compare the prevalence of HIV-related neurocognitive impairment and ADC at the APNAC-10 sites to the published pre-HAART prevalence of these conditions in developed countries
* To compare the prevalence of HIV-related neurocognitive impairment and ADC between the APNAC-10 sites
* To describe the severity of symptoms of patients presenting with symptomatic peripheral sensory neuropathy at the APNAC-10 sites
* To determine the CD4 cell counts, HIV viral loads HIV viral loads and prior ADIs of patients presenting with symptomatic peripheral sensory neuropathy at the APNAC-10 sites
* To determine what proportion of symptomatic peripheral sensory neuropathy may be ascribed to HIV alone, to the use of nucleoside analogues
* To compare the prevalence of symptomatic peripheral sensory neuropathy at the APNAC-10 sites to the published pre-HAART prevalence of these conditions in developed countries
* To compare the prevalence of symptomatic peripheral sensory neuropathy between the APNAC-10 sites
* To determine the prevalence of asymptomatic peripheral neuropathy
* To describe the presenting symptoms and signs of patients presenting with CNS OIs and tumours at the APNAC-10 sites
* To describe the neuroradiological findings of patients presenting with CNS OIs and tumours at the APNAC-10 sites
* To determine the serological, culture and other diagnostic test results of patients presenting with CNS OIs and tumours at the APNAC-10 sites
* To determine the CD4 cell counts, HIV viral loads and prior ADIs of patients presenting with CNS OIs and tumours at the APNAC-10 sites
* To compare the prevalence of CNS OIs and tumours at the APNAC-10 sites to the published pre-HAART prevalence of these conditions in developed countries
* To compare the prevalence of CNS OIs and tumours between the APNAC-10 sites

ELIGIBILITY:
Inclusion Criteria:

* Patients are HIV infected
* Patients are eighteen years or older

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 600
Dates: Start 2005-06

CONTACTS AND LOCATIONS:
Overall Officials: Edwina Wright, Dr, Principal Investigator — The Alfred
Locations (1):
- Alfred Hospital, Melbourne, Victoria, Australia